CLINICAL TRIAL: NCT05781490
Title: An Uncontrolled, Single Centre, Healthy Volunteer, Phase II Proof-of-concept Trial Investigating MR-enterography Image Quality of Lumentin® 44, a New Egg Albumen Based Oral Small Bowel Filling Contrast Agent.
Brief Title: A Healthy Volunteer Trial Investigating MR-enterography Image Quality of Lumentin® 44
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lument AB (Industry)
Collaborators: Q Clinical Research AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LUMRIS-001; 2022-002193-84 (EudraCT Number)
Record Dates: First submitted 2023-02-09; First posted 2023-03-23 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumentin® 44 (Experimental): Lumentin® 44 Powder for oral foam
  Interventions: Drug: Lumentin® 44 Powder for oral foam

INTERVENTIONS:
Drug: Lumentin® 44 Powder for oral foam — Lumentin® 44 is a foam for oral use.

SUMMARY:
A healthy volunteer, open, PoC single center trial investigating a new oral contrast agent for use in combination of MR examination of the abdomen and pelvis.

The main purpose of the trial is to evaluate if Lumentin® 44 used as a bowel filling agent in MRE examination generates images with acceptable diagnostic quality.

In addition, the plasma electrolytes concentration levels, including, potassium, sodium, phosphate, and calcium, as well as ionized calcium will be evaluated over a 24 hour time period after intake of Lumentin.

DETAILED DESCRIPTION:
This is an uncontrolled, single centre phase II trial. Enrolled HVs (n=10) will undergo Gd-enhanced MRE after oral intake of Lumentin® 44.

Interested HVs will be identified primarily among medical students at the medical hospitals at Malmö and Lund. Posters will be placed at the departments and invitation letters will be handed out.

The HVs interested in participating will be invited to attend a pre-screening visit where their suitability based on age and health status will be assessed. Fifteen HVs who fulfil the pre-screening criteria and are interested in participating will be asked to attend a screening visit at the clinic and if eligible for the trial they will then visit the clinic for the MRE assessment within 1-2 weeks.

Only the initial 10 of the eligible HVs will be asked to come for the MRE examination and the remaining eligible subjects will be asked to stand by in case any of the 10 subjects are unable to come or cannot undergo the examination.

HVs will be asked to fast for 6 hours prior to the examination on the day of the MRE examination. Small amount of clear liquid is allowed up to 2 decilitres. Prior to MRE, Lumentin® 44 will be provided to them in volumes of up to 1,500 mL and at least 1,100 mL of Lumentin® 44 must be drunk. The subjects will be asked to drink the solutions of oral contrast agent within 45 minutes to 1 hour.

Subjects not able to drink at least 1.1 L of Lumentin® 44 will be withdrawn from the trial.

Prior to the intake of Lumentin® 44, an IV antecubital cannula will be placed and used for blood sampling and administration of gadolinium (Gd) contrast agent during the MRE assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers of either gender at least 18 years at the time of signing the informed consent.
2. Females must either present a negative pregnancy test or be surgically sterile (hysterectomy or tubal ligation) or postmenopausal (i.e., experienced 12 consecutive months without menstruation).
3. Following verbal and written information about the trial, the subject must provide signed and dated informed consent before any trial related activity is carried out.

Exclusion Criteria:

1. GFR below 60 ml/min/1.73 sqm body surface. All subjects will have a plasma creatinine taken at screening for calculation of eGFR.
2. History of drug related reaction to gadolinium contrast agents.
3. Have had gadolinium injection during the last 4 weeks.
4. Claustrophobia not coping with MRE examination.
5. Metal objects and medical devices in the body not judged by the investigator to be compatible with MRE.
6. Hypersensitivity to Buscopan® (Butylhyoscopin).
7. Having swallowing difficulties.
8. Known allergy to egg albumen.
9. Known sensitivity to any of the components of the investigational product.
10. Clinical suspicion of ongoing disease by the investigator.
11. Being, in the opinion of the investigator, unlikely to comply with the clinical trial protocol.
12. Previously randomized to participate in this trial.
13. Participating in or having participated in another clinical trial within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Leander, Principal Investigator — PeritusClinic
Locations (1):
- PeritusClinic, Lund, Skåne County, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumentin® 44
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 10

OUTCOME MEASURES:

1. Primary Outcome: Visual Evaluation of MRE Images - Motility
Description: Motility: MRE examinations with Lumentin® 44 will be scored with respect to motility status based on a 5-graded scale, as follows:
  1. No motility could be assessed
  2. Motility is assessed to some degree but less good than conventional MRE
  3. Motility is assessed to same degree as conventional MRE
  4. Motility is assessed somewhat better than conventional MRE
  5. Motility is assessed better than conventional MRE Motility should be evaluated as a whole in the specific cine- sequences and resulting in one ordinal score 1-5. A high score indicate a better outcome.
Time Frame: Day 1
Population: All MRE images will be evaluated by one expert radiologist. Only one assessment of each MRE examination will be performed
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  No motility could be assessed | 0
  Motility is assessed to some degree but less good than conventional MRE | 6
  Motility is assessed to same degree as conventional MRE | 4
  Motility is assessed somewhat better than conventional MRE | 0
  Motility is assessed better than conventional MRE | 0

2. Primary Outcome: Visual Evaluation of MRE Images -Artefacts
Description: Artefacts: MRE examinations with Lumentin® 44 will be scored with respect to artefacts based on a 5-graded scale, as follows:
  1. Severe deteriorating artefacts in the interface between the lumen and wall
  2. Disturbing artefacts in the interface between the lumen and wall less good compared to conventional MRE
  3. Medium artefacts in the interface between the lumen and wall, same as for conventional MRE
  4. Small artefacts that give minimal bright edges in the interface between the lumen and wall, somewhat better than conventional MRE
  5. No artefacts and better than conventional MRE Artefacts should be evaluated as a whole in all sequences and resulting in one ordinal score 1-5. A high score indicate a better outcome.
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Severe deteriorating artefacts in the interface between the lumen and wall | 0
  Disturbing artefacts in the interface between lumen and wall less good compared to conventional MRE | 5
  Medium artefacts in the interface between the lumen and wall, same as for conventional MRE | 5
  Small artefacts, minimal bright edges in the interface between lumen/wall, somewhat better than MRE | 0
  No artefacts and better than conventional MRE | 0

3. Primary Outcome: Visual Evaluation of MRE Images -Mucosal Evaluation
Description: Mucosal evaluation: MRE examinations with Lumentin® 44 will be scored with respect to mucosal status based on a 5-graded scale, as follows:
  1. No mucosal folds are seen
  2. Some small mucosal folds can be discriminated
  3. Mucosal folds can be discriminated, same as for conventional MRE
  4. Small mucosal folds can be discriminated, somewhat better than for conventional MRE
  5. Mucosal folds are seen in detail and better than conventional MRE Mucosal evaluation a) coronal and b) axial T1 gradient-echo with Gd should be done and resulting in one ordinal score 1-5. A high score indicate a better outcome.
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  No mucosal folds are seen | 0
  Some small mucosal folds can be discriminated | 6
  Mucosal folds can be discriminated, same as for conventional MRE | 4
  Small mucosal folds can be discriminated, somewhat better than for conventional MRE | 0
  Mucosal folds are seen in detail and better than conventional MRE | 0

4. Primary Outcome: Visual Evaluation of MRE Images -Overall Diagnostic Impression
Description: Overall diagnostic impression: MRE examinations with Lumentin® 44 will be graded for global quality of the information obtained with special reference to diagnostic purposes, as follows:
  1. Poor diagnostic quality
  2. Medium diagnostic quality, below conventional MRE
  3. Good diagnostic quality, same as for conventional MRE
  4. Very good diagnostic quality, somewhat better than conventional MRE
  5. Excellent diagnostic quality, better than conventional MRE The quality of the whole examination and what the impression is for using the examination for diagnostic purposes will be graded on a scale 1-5. A high score indicate a better outcome.
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Poor diagnostic quality | 0
  Medium diagnostic quality, below conventional MRE | 7
  Good diagnostic quality, same as for conventional MRE | 3
  Very good diagnostic quality, somewhat better than conventional MRE | 0
  Excellent diagnostic quality, better than conventional MRE | 0

5. Secondary Outcome: Concentration of Plasma Sodium
Description: Concentration of plasma sodium levels over time
Time Frame: Blood samples will be drawn at baseline just before intake of contrast agent (T0h), and then at 1 hour (T1h), 2 hours (T2h), 4 hours (T4h), 6 hours (T6h), 8 hours (T8h) and at 24 hours (T24h)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
mmol/L
  T0h | 139.70 (1.57)
  T1h | 139.90 (1.20)
  T2h | 140.30 (2.00)
  T4h | 146.60 (1.58)
  T6h | 140.70 (1.83)
  T8h | 140.30 (1.57)
  T24h | 139.80 (1.81)

6. Secondary Outcome: Concentration of Plasma Potassium
Description: Concentration of plasma potassium levels over time
Time Frame: as for outcome 5
Population: Blood samples at various time points could not be analysed due to error in handling of samples.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
mmol/L
  T0h: number analyzed (Participants) | 8
  T0h | 4.04 (0.22)
  T1h | 4.47 (0.24)
  T2h | 4.35 (0.24)
  T4h | 4.16 (0.20)
  T6h: number analyzed (Participants) | 7
  T6h | 4.14 (0.15)
  T8h: number analyzed (Participants) | 8
  T8h | 4.08 (0.17)
  T24h: number analyzed (Participants) | 9
  T24h | 4.10 (0.27)

7. Secondary Outcome: Concentration of Plasma Phosphate
Description: Concentration of plasma phosphate levels over time
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
mmol/L
  T0h | 1.05 (0.31)
  T1h | 1.22 (0.26)
  T2h | 1.35 (0.28)
  T4h | 1.32 (0.27)
  T6h | 1.31 (0.21)
  T8h | 1.32 (0.18)
  T24 | 1.04 (0.38)

8. Secondary Outcome: Concentration of Serum Ionized Calcium
Description: Concentration of serum ionized calcium levels over time
Time Frame: as for outcome 5
Population: Blood samples at various time points could not be analysed due to error in handling of samples.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
mmol/L
  T0h: number analyzed (Participants) | 8
  T0h | 1.28 (0.03)
  T1h: number analyzed (Participants) | 5
  T1h | 1.26 (0.03)
  T2h: number analyzed (Participants) | 5
  T2h | 1.24 (0.04)
  T4h: number analyzed (Participants) | 7
  T4h | 1.26 (0.03)
  T6h: number analyzed (Participants) | 7
  T6h | 1.24 (0.04)
  T8h: number analyzed (Participants) | 7
  T8h | 1.23 (0.02)
  T24h: number analyzed (Participants) | 7
  T24h | 1.28 (0.05)

9. Secondary Outcome: Bowel Filling Properties: Extension/Duodenum
Description: Bowel filling properties: Extension and distension will be evaluated in each of five selected sub-segments of the small bowel. All images will be evaluated by the investigator with respect to how well the small bowel is filled from the bowel through to the terminal ileum (extension) and how well it is distended (distension) by Lumentin® 44. The small bowel will be divided in duodenum, jejunum, proximal ileum, distal ileum and terminal ileum. Both variables will be judged on a scale from 1 to 5, as follows:
  * Extension: 1 is no filling and 5 is filled completely
  * Distension of the segment of small bowel: 1 is no distension and 5 is optimal distension
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Extension/duodenum, Score 1 | 0
  Extension/duodenum, Score 2 | 0
  Extension/duodenum, Score 3 | 0
  Extension/duodenum, Score 4 | 0
  Extension/duodenum, Score 5 | 10

10. Secondary Outcome: Bowel Filling Properties: Extension/Jejunum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Extension/jejunum, score 1 | 0
  Extension/jejunum, score 2 | 0
  Extension/jejunum, score 3 | 0
  Extension/jejunum, score 4 | 0
  Extension/jejunum, score 5 | 10

11. Secondary Outcome: Bowel Filling Properties: Extension/Proximal Ileum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Extension/proximal ileum, score 1 | 0
  Extension/proximal ileum, score 2 | 0
  Extension/proximal ileum, score 3 | 1
  Extension/proximal ileum, score 4 | 0
  Extension/proximal ileum, score 5 | 9

12. Secondary Outcome: Bowel Filling Properties: Extension/Distal Ileum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Extension/Distal ileum, score 1 | 1
  Extension/Distal ileum, score 2 | 0
  Extension/Distal ileum, score 3 | 0
  Extension/Distal ileum, score 4 | 0
  Extension/Distal ileum, score 5 | 9

13. Secondary Outcome: Bowel Filling Properties: Extension/Terminal Ileum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Extension/terminal ileum, score 1 | 3
  Extension/terminal ileum, score 2 | 0
  Extension/terminal ileum, score 3 | 0
  Extension/terminal ileum, score 4 | 0
  Extension/terminal ileum, score 5 | 7

14. Secondary Outcome: Bowel Filling Properties: Distension/Duodenum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Distension/duodenum, Score 1 | 0
  Distension/duodenum, Score 2 | 0
  Distension/duodenum, Score 3 | 2
  Distension/duodenum, Score 4 | 5
  Distension/duodenum, Score 5 | 3

15. Secondary Outcome: Bowel Filling Properties: Distension/Jejunum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Distension/jejunum, Score 1 | 0
  Distension/jejunum, Score 2 | 0
  Distension/jejunum, Score 3 | 5
  Distension/jejunum, Score 4 | 5
  Distension/jejunum, Score 5 | 0

16. Secondary Outcome: Bowel Filling Properties: Distension/Proximal Ileum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Distension/proximal ileum, score 1 | 0
  Distension/proximal ileum, score 2 | 0
  Distension/proximal ileum, score 3 | 1
  Distension/proximal ileum, score 4 | 3
  Distension/proximal ileum, score 5 | 6

17. Secondary Outcome: Bowel Filling Properties: Distension/Distal Ileum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Distension/distal ileum, score 1 | 1
  Distension/distal ileum, score 2 | 0
  Distension/distal ileum, score 3 | 0
  Distension/distal ileum, score 4 | 1
  Distension/distal ileum, score 5 | 8

18. Secondary Outcome: Bowel Filling Properties: Distension/Terminal Ileum
Description: as for outcome 9
Time Frame: MR examination, Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lumentin® 44
Number analyzed (Participants) | 10
Participants
  Distension/terminal ileum, score 1 | 3
  Distension/terminal ileum, score 2 | 0
  Distension/terminal ileum, score 3 | 0
  Distension/terminal ileum, score 4 | 3
  Distension/terminal ileum, score 5 | 4

ADVERSE EVENTS:
Time Frame: From start of intake of study medication and 2 days after treatment. Trial subjects were in the trial between 23 JAN 2023 and 17 FEB 2023
Arm/Group | Lumentin® 44
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumentin® 44 (N=10)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT05781490/Prot_SAP_000.pdf